CLINICAL TRIAL: NCT06720961
Title: Unveiling the Microbial Impact on Intestinal Fibrosis and the Associated Immune Microenvironment: New Insights for the Pathogenesis and Treatment of Crohn's Disease-associated Complications
Brief Title: The Microbial Impact on Intestinal Fibrosis and the Associated Immune Microenvironment in Crohn's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: University of Florence (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Ministero dell'Istruzione, dell'Università e della Ricerca (Unknown); Università Vita-Salute San Raffaele (MI) (Unknown)
Responsible Party: Principal Investigator, Silvio Danese, Professor, IRCCS San Raffaele
Other Study IDs: PRIN-2022RKE4L; Bando MUR 2022 PRIN-2022RKE4L (Other Grant/Funding Number: Ministero dell'Università e della Ricerca (MUR))
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease (CD)
Keywords: Crohn Disease; Fibrosis; Dysbiosis; Microbiota; Fibrostenosis
MeSH Terms: conditions — Crohn Disease; Fibrosis; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bioptic surgical specimens will be collected according to standard of care and, for the study, we will use leftover material after pathologist analysis.
  One week before the surgery the collection of fecal material from CD and from non-IBD patients will be performed ad hoc for clinical research purposes of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD Patients: CD patients with established diagnosis and additionally classified according to 3 stages: B1 (more inflammatory, non-stricturing), B2 (stricturing, non-penetrating) and B3 (stricturing and penetrating). Patients will be stratified on the basis of CT, MRI or ultrasound analysis (stratification already known before surgery)
  Interventions: Procedure: Collection of surgical specimen; Procedure: Collection of stool sample
- Non-IBD Patients: Patients with other pathologies but not affected by IBD according to the previously reported clinical and endoscopic evaluation criteria (ex. diverticulitis)
  Interventions: Procedure: Collection of surgical specimen; Procedure: Collection of stool sample

INTERVENTIONS:
Procedure: Collection of surgical specimen — Specimens of CD patients and non-IBD related patients will be collected during the surgery performed for clinical practice, without other risks for the patients, since we will use only leftover material after pathologist analysis. All of the collected surgical samples will be used for this project and, for this reason, they will not be conserved after the research period. Any residual samples will be destroyed.
Procedure: Collection of stool sample — One week before the surgery to remove the stricture, fecal samples from CD patients belonging to B1, B2, B3 groups will be collected. They will be used for the exploratory objective. All of the collected fecal samples will be used for this project and, for this reason, they will not be conserved after the research period. Any residual samples will be destroyed.

SUMMARY:
The goal of this study is to find out if there is a direct connection between an imbalance of gut bacteria and the development of scar tissue in the gut by identifying important bacterial proteins found in scarred gut tissue. Our aim is to identify which types of cells and biological processes are affected by these bacterial proteins in people with Crohn's Disease. We will also study how these bacterial proteins cause changes in 3D models of gut fibrosis.

DETAILED DESCRIPTION:
More than 50% of CD patients develop a penetrating disease or stenosis due to fibrostenosis, which in most cases requires surgery, as no effective therapies have yet been found. The disease leads to both structural and functional alterations of the intestinal mucosa. Although the functional alteration of the mucosa is mainly caused by the continuous tissue damage that occurs during the chronic inflammation associated with CD, recent studies have suggested that the fibrosis associated with CD may be driven by triggering factors independent of inflammation, such as dysbiosis of the microbiota. Our proposal aims to establish the causal link between gut dysbiosis and fibrosis by studying the role of key bacterial proteins present in fibrotic gut tissue.

This project will ultimately offer new molecular targets for the development of possible tailor-made antifibrotic treatments, with likely benefits for healthcare, as it will facilitate the management of severe CD, avoiding surgery and reducing SSN costs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 and <70 years
* Patients able to autonomously sign the informed consent
* Non pregnant or breastfeeding patients
* For CD patients: CD patients with established diagnosis and additionally classified according to 3 stages: B1 (more inflammatory, non-stricturing), B2 (stricturing, non-penetrating) and B3 (stricturing and penetrating). Patients will be stratified on the basis of CT, MRI or ultrasound analysis (stratification already known before surgery)
* For non-IBD patients: patients with other pathologies but not affected by IBD according to the previously reported clinical and endoscopic evaluation criteria (ex. diverticulitis)

Exclusion Criteria:

* Patients <18 years or > 70 years
* Pregnant or breastfeeding patients
* For CD Patients: Subjects with CD who do not meet evaluation criteria described above
* For non-IBD patients: Patients undergoing anti-inflammatory and/or immunosuppressive treatments for IBD-related diseases

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll 15 CD patients and 5 patients without IBD-related diseases (ex. diverticulitis) undergoing surgery according to the normal clinical practice for a total of 20 patients as following:
  - 15 patients with CD (5 patients/stage: B1 (more inflammatory, non-structuring), B2 (structuring, non-penetrating) and B3 (structuring and penetrating).
  Patients will be stratified according to CT, MRI or ultrasound analysis (stratification already known before surgery)
  - 5 patients without IBD-related diseases (e.g. diverticulitis)
  All patients will be recruited only from San Raffaele Hospital (OSR). The participation is voluntary and the patient is allowed to refuse further participation in the protocol whenever he/she wants.
  Participation in the study will not change the diagnostic-therapeutic treatment that patients undergo following the clinical practice, since patients will continue to be treated in accordance with clinical practice regardless of the results of this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To identify the cellular subtypes and molecular pathways impacted by the specific bacterial factors during CD-associated fibrosis. | Experiments and analysis: 11th to 36th month
  Control subjects' and CD-derived surgical specimens will be processed to obtain a cell suspension, that will be frozen and stored for the subsequent cell sorting. Frozen CD and healthy cell suspensions will be then thawed and undergo FACS for specific cell markers (CD31 for endothelial cells, EpCam for epithelial cells, CD90 for fibroblasts, CD45 for leukocytes, including CD4 and CD8 for T cells, CD20 for B cells, CD14 and CD163 for macrophages (MΦ), CD11b and c for dendritic cells (DCs). Single-cell populations will undergo library preparation and will be analyzed by ribo-minus RNAseq at 30M reads of depth.
  Metatranscriptomics for profiling the microbial composition, as well as the transcriptomics to determine both the differential gene expression (DGE) and the Gene Set Enrichment Analysis (GSEA), will be performed.

SECONDARY OUTCOMES:
To unravel the cellular and molecular mechanisms and dynamics induced by the bacterial factors in 3D models of intestinal fibrosis | Experiments and analysis: 11th to 36th month
  We will isolate and sequence RNA of specific cellular subtypes from the phenotype B1, B2, and B3 of fibrotic CD tissues and healthy non-IBD tissues.
  We will profile the microbial composition by Metatranscriptomics as well as we will determine both the differential gene expression (DGE) and the Gene Set Enrichment Analysis (GSEA) through transcriptomics.
  Moreover, to identify the cellular type(s) where bacterial proteins will be expected to exert the most prominent pro-fibrotic effects, we will set up the transwell-based experimental platform by plating epithelial cells (organoids) and/or endothelial cells, and/or fibroblasts in the upper chamber of the transwell, while lamina propria mononuclear cells (LPMCs) will be plated in the lower chamber

OTHER OUTCOMES:
To validate in vitro results in an animal model by assessing the role of microbial factors in inducing fibrosis in an entire organism. Moreover, we will provide a possible therapeutic approach with strong clinical implications in the future | Experiments on in-vivo models: 13th to 24th month
  To evaluate the efficacy of nanomedicine therapy in inhibiting the deleterious processes induced by bacterial factors by exploiting in vivo models that recapitulate CD-associated fibrosis.
  We will evaluate the pro-fibrotic potential of specific bacterial factors during experimental intestinal fibrosis, testing a possible treatment through the liposome-mediated inhibition of bacterial factor-induced mechanisms. For this. purpose, fecal samples collected from patients will be handled and processed for analysis in our Lab and will then be shipped to UO2 for in vivo studies

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, PhD-MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided